CLINICAL TRIAL: NCT03161327
Title: Positive Predictive Value of Digital Ankle Brachial Index (ABI) as a Screening Tool in Detecting Peripheral Arterial Disease: A Single Center, Prospective Clinical Trial
Brief Title: Digital Ankle Brachial Index (ABI) as a Screening Tool in Detecting Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Keith Pereira, MD:, Assistant Professor, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 28225
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Peripheral Artery Disease; Amputation; Smoking; Diabetes; Hypercholesterolemia; Hypertension
Keywords: ankle brachial index; peripheral arterial disease
MeSH Terms: conditions — Peripheral Arterial Disease; Smoking; Diabetes Mellitus; Hypercholesterolemia; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ABI (Other): ABI will be performed in patient
  Interventions: Device: ABI using QuantaFlo™

INTERVENTIONS:
Device: ABI using QuantaFlo™ — Perform Digital ABI:
  * Will be performed by the nurse/medical assistant with training to perform this test
  * The patient will be placed in the supine position, with the arms and legs at the same level as the heart, for a minimum of 5 minutes before measurement.
  * The optical sensor (similar to a pulse oximeter) will be placed sequentially in the fingers of the hands and feet: Right and left hand fingers and then right and left feet toes.
  * Usually each digit takes about 15 seconds to obtain a waveform
  * At the end of 60 seconds, an automated digital ABI will be generated.
  Clinical course: If based on Screening questionnaire and digital ABI, I. Patient is diagnosed with PAD- the referring physician and patient will receive a phone call about the same. He/ she will then be advised any further testing/ referral to IR clinic.
  II. There is no evidence of PAD- no further action will be taken. The patient will be informed of the same.

SUMMARY:
Peripheral artery disease (PAD) affects 8-18 million in the US and is an economic burden, currently estimated to be greater than cancer and heart disease. Older age (> 65 years), smoking, diabetes and kidney diseases are some risk factors associated with PAD and are known to have increased morbidity and mortality.Early detection is critical for mitigating PAD progression. Ankle-brachial index (ABI) testing is recommended by the US Preventative Services Task Force as an affordable and effective screening tool for evaluating PAD risk.

QuantaFlo™ (Semler Scientific, Inc.) is a novel, noninvasive, 510K FDA approved digital device that is used as a screening tool to measure ABI of patients at risk of PAD. This single center prospective clinical trial will evaluate the sensitivity and specificity of digital ABI in detecting PAD using color Doppler ultrasound and 'gold standard' angiography as reference. Specifically in patient undergoing dialysis and who cannot undergo ABI using pressure cuffs dialysis grafts/ fistulae in the arms, we will evaluate the value of digital ABI in detecting PAD.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) affects 8-18 million in the US and is an economic burden, currently estimated to be greater than cancer and heart disease. Older age (> 65 years), smoking, diabetes and kidney diseases are some risk factors associated with PAD and are known to have increased morbidity and mortality. PAD progression directly results in claudication, impaired walking, and amputation. Amputation is not benign - impacts are physical and emotional. Recovery from amputation involves long-term rehabilitation. The American Heart Association (AHA) in 2016 guidelines suggests an algorithm for diagnosis and management of PAD. They recommend a collaborative multidisciplinary team approach between the primary care physician and specialists including; a diabetologists/ endocrinologist, smoking cessation expert, hypertension and lipid specialist, interventional radiologist, vascular surgeon, orthopedist, neurologist, wound healing expert, and/or others for 'the greatest chance of providing optimal care for the patient with PAD'.

Early detection is critical for mitigating PAD progression. Ankle-brachial index (ABI) testing is recommended by the US Preventative Services Task Force as an affordable and effective screening tool for evaluating PAD risk. ABI testing is especially useful in primary care settings allowing for earlier diagnosis and treatment. Several ABI methods are used; classically this test uses a device for measuring blood pressure with an inflatable cuff, and blood pressure measurements are taken at the upper arm and the ankle; healthcare providers have used a doppler probe to detect audible systolic pressure signals within the arteries - Doppler ABI. Barriers to implementation include; time required to conduct tests, training and required technical skills. Hence, Doppler-based ABI in primary care has been limited. Recently designed oscillometric (manual or digital with automatic electronic calculation of blood pressure) and photophlethysmographic devices are now available. However current guidelines do not endorse the use of these newer devices but recommend the hand-held doppler technique.

Digital ABI is noninvasive, automated ABI using pulsatile blood volume changes - plethysmography, irrespective of vessel compressibility. The QuantaFlo™ (Semler Scientific, Inc.) is an innovative, 510K FDA approved device that provides bilateral, non-invasive physiologic studies of upper and lower extremity arteries using volume plethysmography of the posterior tibial and anterior tibial/dorsalis pedis arterial distributions. QuantaFlo™ uses an optical sensor attached onto a digit in the hand and feet to assess extremity blood volume. It then displays a signal, directly related to blood volume, on a Volume Plethysmography Chart used to calculate PAD probability. This test is easy to use and portable, delivering fast, accurate results in ~5 minutes; an attractive option in primary care settings. While maintaining accuracy, results comparing digital methods to Doppler show concordance above 90%. The American Medical Association (AMA) concluded, "Evaluation of the digits in both legs with volume plethysmography is appropriate for this code provided that an ankle/brachial index (ABI) be performed." QuantaFlo™ meets both of these standards.

ABI ≤ 0.9 has been used as the criterion for diagnosing PAD based on ACC/AHA guidelines for the management of patients with PAD ; the cutoff value of ABPI ≤0.9 it has been reported that the sensitivity of diagnosing PAD was 83% to 85% and a specificity of 95% to 100% [5]. ABI has been validated against lower extremity contrast angiography obtaining high sensitivity (85%-95%) and specificity (90%-100%), for diagnosing PAD . Many studies have reported more than 95% of sensitivity and specificity of colour duplex ultrasound scan in detecting a significant stenosis of the arteries .

QuantaFlo™ (Semler Scientific, Inc.) is a novel, noninvasive, 510K FDA approved digital device that is used as a screening tool to measure ABI of patients at risk of PAD. This single center prospective clinical trial will evaluate the sensitivity and specificity of digital ABI in detecting PAD using color Doppler ultrasound and 'gold standard' angiography as reference. Specifically in patient undergoing dialysis and who cannot undergo ABI using pressure cuffs dialysis grafts/ fistulae in the arms, we will evaluate the value of digital ABI in detecting PAD.

ELIGIBILITY:
Inclusion Criteria:

Answering yes to any of the following questions on the clinical screening questionnaire:

* Are you 65 years or older?
* Have you ever smoked?
* Do you have diabetes?
* Do you have high blood pressure or take medication for high blood pressure?
* Do you have high cholesterol, or take medication for high cholesterol?
* Have you previously had a stroke?
* Do you have heart disease?
* Do you experience any pain at rest in your lower legs or feet?
* Do you have discomfort (aching, fatigue, tingling, cramping or pain) when you walk, which is relieved by rest? Does the pain go away within 10 minutes after stopping?
* Are your toes or feet pale, discolored, or bluish?
* Do you have an infection, skin wound, or ulcer on your feet or toes?

Exclusion Criteria:

* Not meeting the above criteria.
* Previously screened with ABI in past 12 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Pereira, MD, Principal Investigator — Saint Louis University Hospital
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited patients from various clinics presenting for appointments not necessarily related to PAD. Patients were asked to complete a screening questionnaire. 1791 patients completed the questionnaire. Patients giving any yes responses were asked if they wanted to participate in the study.
Pre-assignment Details: Of the 1791 patients who completed the survey, 238 enrolled in the study (gave consent and completed digital ABI screening).
Groups:
- Patients at Risk for PAD: For those who screened positive by the questionnaire, and signed consent, a digital ABI was performed using QuantaFlo™. For subjects with PAD the referring physician and patient will receive a phone call about the same. He/ she will then be advised any further testing/ referral to IR clinic. For subjects with no evidence of PAD, subject will be informed of results, and no further action taken.
Period: Overall Study
Arm/Group | Patients at Risk for PAD
Started | 238
Completed | 238
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 238-missing 32 data sheets = 206
Arm/Group | Patients at Risk for PAD
Number analyzed (Participants) | 206
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 125
  >=65 years | 81
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: ABI severe, mod and mild risk categories are made up of subjects within the overall at risk for PAD population. These categories are based on ABI results of that population.
  years
    All patients at risk for PAD | 59.9 (13.1)
    ABI severe risk: number analyzed (Participants) | 10
    ABI severe risk | 68.2 (8.5)
    ABI moderate risk: number analyzed (Participants) | 15
    ABI moderate risk | 65.6 (9.2)
    ABI mild risk: number analyzed (Participants) | 19
    ABI mild risk | 67.1 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: ABI severe, mod and mild risk categories are made up of subjects within the overall at risk for PAD population. These categories are based on ABI results of that population.
  Participants
    ABI severe risk: number analyzed (Participants) | 10
    ABI severe risk: Female | 6
    ABI severe risk: Male | 4
    ABI moderate risk: number analyzed (Participants) | 15
    ABI moderate risk: Female | 9
    ABI moderate risk: Male | 6
    ABI mild risk: number analyzed (Participants) | 19
    ABI mild risk: Female | 16
    ABI mild risk: Male | 3
    All patients at risk for PAD: Female | 128
    All patients at risk for PAD: Male | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
diabetic [Count of Participants; unit: Participants]
  Pateients at risk for PAD | 100
  ABI severe risk | 6
  ABI moderate risk | 11
  ABI mild risk | 11

OUTCOME MEASURES:

1. Primary Outcome: Positive Predictive Value of Digital ABI in Diagnosing PAD
Description: To evaluate the Positive predictive value of digital ABI in diagnosing PAD using color Doppler ultrasound and 'gold standard' angiography as reference.
Time Frame: 3 months
Population: Positive Predictive Value (PPV)
Measure: Count of Participants; unit: Participants
Groups:
- ABI Severe Risk: Those who screened at risk for PAD on questionnaire, had digital ABI performed, and if ABI <0.4 , these were described as severe risk for PAD
- ABI Moderate-mild Risk: Those who screened at risk for PAD on questionnaire, had digital ABI performed, and results were 0.4 to 0.9 , these were at moderate or mild risk for PAD
Arm/Group | ABI Severe Risk | ABI Moderate-mild Risk
Number analyzed (Participants) | 10 | 34
Participants | 8 | 2

ADVERSE EVENTS:
Time Frame: Data was collected over the time of performing the non invasive ABI test. This was for 2 months
Description: Adverse Even (AE) any adverse event occurring at the time of or following time of procedure/ embolization through the remainder of study.
  Serious Adverse Event (SAE):
  * death during the period of protocol defined surveillance
  * persistent or significant disability/incapacity.
  Unanticipated Adverse Event (UAE): any event that could not be reasonably foreseen or had not been previously reported in the product package insert as a potential adverse event related to use of this device
Groups:
- ABIABI Using QuantaFlo™: ABI will be performed in patient
  ABI using QuantaFlo™: Perform Digital ABI:
  * Will be performed by the nurse/medical assistant with training to perform this test
  * The patient will be placed in the supine position, with the arms and legs at the same level as the heart, for a minimum of 5 minutes before measurement.
  * The optical sensor (similar to a pulse oximeter) will be placed sequentially in the fingers of the hands and feet: Right and left hand fingers and then right and left feet toes.
  * Usually each digit takes about 15 seconds to obtain a waveform
  * At the end of 60 seconds, an automated digital ABI will be generated.
  Clinical course: If based on Screening questionnaire and digital ABI, I. Patient is diagnosed with PAD- the referring physician and patient will receive a phone call about the same. He/ she will then be advised any further testing/ referral to IR clinic.
  II. There is no evidence of PAD- no further action will be taken. The patient will be informed
Arm/Group | ABIABI Using QuantaFlo™
All-Cause Mortality (participants affected / at risk) | 0/238
Serious Adverse Events (participants affected / at risk) | 0/238
Other Adverse Events (participants affected / at risk) | 0/238

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT03161327/Prot_SAP_000.pdf